CLINICAL TRIAL: NCT06766695
Title: A Survey Study on the Job Burnout of Chinese Endoscopy Nurses
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 研2024-1312
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Occupational Burnout
Keywords: Occupational burnout; Sleep condition; Chinese endoscopy nurse; Emotional state
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Occupational burnout (burnout) was proposed by American psychologist Herbert Freudenberger in 1974, who it as a syndrome caused by prolonged exposure to workplace stress that is not successfully managed. Subsequently, Maslach et al. believed that occupational burnout refers an excessive physical and mental consumption state of individuals under prolonged work pressure, including emotional exhaustion, depersonalization, and low personal accomplishment. In January 222, the WHO's "International Classification of Diseases, 11th Edition" included "occupational burnout" for the first time, officially recognizing as a disease, considering occupational burnout to be a syndrome caused by prolonged work pressure that is not effectively managed. Compared with other professions, doctors and nurses are higher risk of occupational burnout. Occupational burnout is closely related to the work quality of medical staff, doctor-patient relationship, and mental and physical health. 2022, 47% of 13,000 doctors in the United States experienced occupational burnout. Whether occupational burnout mental and physical health, thereby affecting the quality of medical care, deserves further study. This study plans to use a questionnaire survey method to analyze the status of occupationalout, emotional state, and sleep among nurses in endoscopy centers in mainland China, providing reference for medical staff to take measures to cope with occupational burnout improve mental and physical health, and the quality of medical care.

DETAILED DESCRIPTION:
Occupational burnout (burnout) was proposed by American psychologist Herbert Freudenberger in 1974, who it as a syndrome caused by prolonged exposure to workplace stress that is not successfully managed. Subsequently, Maslach et al. believed that occupational burnout refers an excessive physical and mental consumption state of individuals under prolonged work pressure, including emotional exhaustion, depersonalization, and low personal accomplishment. In January 222, the WHO's "International Classification of Diseases, 11th Edition" included "occupational burnout" for the first time, officially recognizing as a disease, considering occupational burnout to be a syndrome caused by prolonged work pressure that is not effectively managed. Compared with other professions, doctors and nurses are higher risk of occupational burnout. Occupational burnout is closely related to the work quality of medical staff, doctor-patient relationship, and mental and physical health. 2022, 47% of 13,000 doctors in the United States experienced occupational burnout. Whether occupational burnout mental and physical health, thereby affecting the quality of medical care, deserves further study. This study plans to use a questionnaire survey method to analyze the status of occupationalout, emotional state, and sleep among nurses in endoscopy centers in mainland China, providing reference for medical staff to take measures to cope with occupational burnout improve mental and physical health, and the quality of medical care.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in endoscopy centers on the Chinese mainland were selected and completed the questionnaire online after informed consent. Inclusion criteria: ① to cooperate in completing the questionnaire; ② no history of mental illness.

Exclusion Criteria:

* Failed to fill out all the scales effectively.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nurses from endoscopy centers in mainland China were selected and completed the questionnaire online after informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
A Survey Study on the Job Burnout of Chinese Endoscopy Nurses | 2025.1.5-2026.12.30
  article

IPD SHARING:
Plan to Share IPD: No